CLINICAL TRIAL: NCT02436213
Title: Hypoxemia, Dyspnea, and Exercise Tolerance in Patients With Pulmonary Arteriovenous Malformations
Brief Title: Cardiopulmonary Exercise Testing to Evaluate Pulmonary AVMs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLS/22; 11/H0803/9 (Other: National Research Ethics Service, UK)
Record Dates: First submitted 2012-10-16; First posted 2015-05-06 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Arteriovenous Malformations; Hereditary Hemorrhagic Telangiectasia
Keywords: workload; oxygen level; oxygen consumption; breathing reserve; ventilatory efficiency
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Exercise Test; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (Experimental): A group of up to 30 healthy controls will be recruited to have a cardiopulmonary exercise test and a blood test.
  Interventions: Other: Cardiopulmonary exercise test; Procedure: Blood test
- Pulmonary AVM (Experimental): A group of up to 30 pulmonary AVM patients will be recruited to have a cardiopulmonary exercise test, and a blood test.
  Interventions: Other: Cardiopulmonary exercise test; Procedure: Blood test
- HHT but no pulmonary AVM (Experimental): Most patients with pulmonary AVMs have underlying hereditary hemorrhagic telangiectasia (HHT). If there is a difference between pulmonary AVM and control groups that does not correct following embolization of pulmonary AVMs, a group of up to 30 people with HHT but no evidence of pulmonary AVMs will be selected to have a cardiopulmonary exercise test and a blood test.
  Interventions: Other: Cardiopulmonary exercise test; Procedure: Blood test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — On Day 1, subjects will have the test in the Exercise Suite of Hammersmith Hospital, London, UK. They will have painless skin probes placed on their fingers, chest, and legs to monitor heart rate, ECG, blood oxygen levels, and oxygen delivery during the test. Subjects will also be shown how to breathe through a mouthpiece with a nose clip on, and how to indicate on a sliding device whether they feel breathless. They will then start cycling against a very low resistance at a steady speed. As long as they feel comfortable, there will be a gradual increase in work load until they feel they cannot keep going at the same speed. They can also stop sooner for any reason. Afterwards, while they are "cooling down" (within the hour on Day 1), they will fill in a short questionnaire describing how they feel.
Procedure: Blood test — On same day (Day 1), the subject will have 20-30mls of blood (that is, 4-6 teaspoonful) taken for analysis.

SUMMARY:
Pulmonary arteriovenous malformations (PAVMs) are a rare vascular condition affecting the lungs. PAVMs lead to low blood oxygen levels, yet are very well tolerated by patients. This study will examine the exercise capacity of PAVM patients using formal cardiopulmonary exercise tests performed on a stationary bicycle.

DETAILED DESCRIPTION:
It is well known that the lung is the site at which oxygen enters the blood stream, diffusing from the alveolar air sacs into the pulmonary capillaries. This newly oxygenated blood is carried to the heart in the pulmonary veins, then passes into the systemic circulation to provide oxygen to the tissues.

Patients with pulmonary arteriovenous malformations (PAVMs) have abnormal vascular connections between pulmonary arteries and pulmonary veins in the lung. Blood flowing through PAVMs therefore bypasses the oxygenation sites in the pulmonary capillaries. Low blood oxygen levels (hypoxemia) is frequent in PAVM patients but breathlessness (dyspnea) is not. The investigators have shown that dyspnea was not a common presenting complaint in a large UK series, and that there is little correlation between severity of dyspnea in PAVM patients, and blood oxygen levels.

In this study the investigators will address the question "Why are hypoxemic PAVM patients not more dyspneic?"

The investigators will address this by first performing standardised cardiopulmonary exercise testing, as used in the clinic, on age and sex matched patients with PAVMs and healthy controls. Physiological parameters will be compared, to test the null hypothesis that the impact of exercise on PAVM patients' cardiopulmonary systems does not differ to normal controls.

If the expected differences are confirmed, the investigators will examine if there is any difference to normals by re-examining the exercise tolerance of the PAVM cohort after they have had their PAVMs treated by embolization.

Most patients with PAVMs have an underlying hereditary vascular disorder, hereditary haemorrhagic telangiectasia. Assuming the expected differences between PAVM patients and controls are confirmed, the investigators will therefore also examine which pattern HHT patients without PAVMs display. Finally, cellular and molecular methods will be used to dissect mechanistic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Healthy volunteers: no concurrent health reason to avoid exercise
* Pulmonary AVMs: pulmonary AVMs confirmed by CT scan
* Hereditary hemorrhagic telangiectasia without pulmonary AVMs: HHT according to current international consensus criteria, with no evidence of PAVMs on dedicated thoracic CT scan.

Exclusion Criteria:

* Inability to provide informed consent.
* Any known cardiovascular abnormality including a history of syncope (faintness, dizziness, lightheadedness or loss of consciousness due to an abnormality of the cardiovascular system).
* Current respiratory tract infection (eg a cold).
* Pregnancy.
* Claustrophobia or needle phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total body oxygen consumption in mls/min/kg, at peak exercise (VO2 max). | Same day (Day 1), at end of exercise study
  Of the many measurements and derived indices that can be measured during cardiopulmonary exercise testing, the peak consumption of oxygen (VO2 max) is perhaps the best indicator of integrated cardiorespiratory capacity. The principle research question will therefore test the null hypothesis that "The VO2 max does not differ between PAVM patients and age matched healthy controls."

SECONDARY OUTCOMES:
Breathing reserve (%) | Same day (Day 1) at end of exercise test
  We will also test in univariate and multiple regression analyses whether breathing reserve differs between PAVM patients and controls.
Ventilatory efficiency, derived from the VE / CO2 slope (L/min/L/min) | Same day (Day 1), at end of exercise study
  We will also test in univariate and multiple regression analyses whether ventilatory efficiency differs between PAVM patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, Du Cane Rd, London, United Kingdom

REFERENCES:
- [Result] Howard LSGE, Santhirapala V, Murphy K, Mukherjee B, Busbridge M, Tighe HC, Jackson JE, Hughes JMB, Shovlin CL. Cardiopulmonary exercise testing demonstrates maintenance of exercise capacity in patients with hypoxemia and pulmonary arteriovenous malformations. Chest. 2014 Sep;146(3):709-718. doi: 10.1378/chest.13-2988. PMID 24676541
- [Result] Gawecki F, Strangeways T, Amin A, Perks J, McKernan H, Thurainatnam S, Rizvi A, Jackson JE, Santhirapala V, Myers J, Brown J, Howard LSGE, Tighe HC, Shovlin CL. Exercise capacity reflects airflow limitation rather than hypoxaemia in patients with pulmonary arteriovenous malformations. QJM. 2019 May 1;112(5):335-342. doi: 10.1093/qjmed/hcz023. PMID 30657990